CLINICAL TRIAL: NCT03114072
Title: Nightly Light Exposure in Pregnancy: Blue-blocking Glasses as an Intervention to Ease Sleep Disturbances and to Improve Mood
Brief Title: Blocking Blue Light in Pregnancy, Effects on Melatonin Profile and Sleep
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: The Norwegian Competence Center for Sleep Disorders (SOVno) (Unknown); Western Norway University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Randi Liset, Principal Investigator, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016/1394/REK vest
Record Dates: First submitted 2017-03-24; First posted 2017-04-14 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Sleep Disturbance
Keywords: Pregnancy; Blue-blockers; Sleep quality; Melatonin
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Consenting participants will be randomized (by www.randomizer.org) to either intervention/control condition. The intervention- and control glasses will be covered in the same looking wrapping, done by a third person, which will blind the investigator as well.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blue-blocking glasses (Active Comparator): N=30 The Blue-blocking glasses (orange-tinted), which remove more than 99% of the blue wavelengths (wavelengths within the visible spectrum shorter than 530 nm). Luminous transmittance: 50%.
  Interventions: Device: Blue-blocking glasses
- Light grey control glasses (Active Comparator): N=30 Partially blue blocking light grey glasses, blocking only about 50% of blue wavelengths (wavelengths within the visible spectra shorter than 530 nm). Luminous transmittance: 55%.
  Interventions: Device: Light grey control glasses

INTERVENTIONS:
Device: Blue-blocking glasses — Wear the BB-glasses from three hours before bedtime, and if needed to turn on the light, also during the night.
  Other Names: Virtual darkness eyewear, orange glasses
  Arms: Blue-blocking glasses
Device: Light grey control glasses — Wear the light grey glasses from three hours before bedtime, and if needed to turn on the light, also during the night.
  Other Names: Grey sunglasses
  Arms: Light grey control glasses

SUMMARY:
Sleep disturbances are common in pregnancy, and the incidence increases during the third trimester. Light and specially the blue wavelengths of light, is affecting sleep and the circadian rhythm. The main aim of this randomized controlled study is to investigate the effect of Blue-blocking glasses (BB-glasses) used in the evening and night on sleep and mood in pregnant women in the third trimester. The outcome measures assess sleep variables, alertness, melatonin level, sleepiness (subjectively), mood and symptoms of anxiety and depression. In addition we want to measure the pregnancy related sleep problems, alcohol intake, physical activity and perceives stress in the study population, and the association with daily/nightly light exposure.

DETAILED DESCRIPTION:
Several hormonal and mechanical influences can cause insomnia in pregnancy, and insomnia has been reported by 62% of pregnant women, a number that is significantly higher than found in the general population (10-15%). Disrupted sleep among pregnant women also includes nocturia (a frequent need to get up and urinate at night), dyspnea (shortness of breath), nasal congestion, muscular aches and pelvic pains, fetal activity, leg cramps as well as reflux.

Artificial light in the evening and during the night increases alertness, disturbs sleep, shifts the timing of the circadian clock and impairs the brains' restorative slow waves during deep sleep. Recent studies have however shown that use of BB-glasses in the evening improves sleep quality (subjectively reported) among persons with insomnia, and prevent alertness caused by blue-light emitting screens which are part of devices such as smart-phones and tablets.

This project will contribute with new knowledge on how filtering nightly light exposure in pregnant women in their third trimester affects their sleep and mood. Importantly, the project initiates new research on a potential non-pharmacological treatment of sleep disturbances by blocking blue wavelengths of light in the evening and during nocturnal awakenings. Blue light is known to increase alertness through a recently described retinal receptor; the intrinsically photoresponsive retinal ganglion cell (IpRGC), specialized for detecting daytime light signal. This project is highly innovative and may have significant practical implications Due to the variety of aims and outcome measures, we plan to present the outcomes in separate articles.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous women
* expecting one child
* being in the third trimester of a normal pregnancy
* able to wear an actigraph during daytime and nighttime
* able to fill out a questionnaire in Norwegian

Exclusion Criteria:

* somatic or psychiatric disorders
* fever and other health conditions affecting sleep
* working at night during the study protocol

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant human beings are female.
Enrollment: 60 (Estimated)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Sleep diary | 3 weeks in the third trimester of pregnancy, mainly gestational week 28-31
  Daily subjective estimates of sleep variables, and will be assessed every morning.
Change in motor activity measured by using Actigraphy. | 3 weeks in the third trimester of pregnancy, mainly gestational week 28-31
  Objective measure by Actiwatch Spectrum from Philips Respironics. The participants will use the Actiwatch for the whole study period of three weeks.
Melatonin level | 3 weeks in the third trimester of pregnancy, mainly gestational week 28-31
  Measured by saliva samples.

SECONDARY OUTCOMES:
Bergen Insomnia Scale (BIS) | 3 weeks in the third trimester of pregnancy, mainly gestational week 28-31
  The BIS measure subjective symptoms of insomnia during the previous week, and will be assessed at day 1 and day 21 of the study period.
Karolinska Sleepiness Scale (KSS) | 3 weeks in the third trimester of pregnancy, mainly gestational week 28-31
  Measure subjective sleepiness just prior to turning the lights off, and will be assessed every evening in the study period.
Evening activation | 3 weeks in the third trimester of pregnancy, mainly gestational week 28-31
  Measured subjectively by the Pre-Sleep Arousal Scale (PSAS).
Sleepiness (subjectively) | 3 weeks in the third trimester of pregnancy, mainly gestational week 28-31
  Measured by the Epworth Sleepiness Scale (ESS).
Mood | 3 weeks in the third trimester of pregnancy, mainly gestational week 28-31
  Measured by the self-report forms Positive and Negative Affect Schedule.
The Beck Anxiety Inventory (BAI) | 3 weeks in the third trimester of pregnancy, mainly gestational week 28-31
  Measure subjective symptoms of anxiety, and will be assessed at day 1 and day 21 of the study period.
The Beck Depression Inventory-II (BAI-II) | 3 weeks in the third trimester of pregnancy, mainly gestational week 28-31
  Measure subjective symptoms of depression during the last week, and will be assessed at day 1 and day 21 of the study period.
Common pregnancy complaints Questionnaire | 3 weeks in the third trimester of pregnancy, mainly gestational week 28-31
  Measure subjective complaints during the last night, assessed every morning of the study period.
Cortisol level | 3 weeks in the third trimester of pregnancy, mainly gestational week 28-31
  Measured by saliva samples, assessed at day 7 and day 21 of the study period.
Alpha Amylase level | 3 weeks in the third trimester of pregnancy, mainly gestational week 28-31
  Measured by saliva samples, assessed at day 7 and day 21 of the study period

CONTACTS AND LOCATIONS:
Overall Officials: Randi Liset, PhD, Principal Investigator — University of Bergen
Locations (1):
- Randi Liset, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbott SM, Attarian H, Zee PC. Sleep disorders in perinatal women. Best Pract Res Clin Obstet Gynaecol. 2014 Jan;28(1):159-68. doi: 10.1016/j.bpobgyn.2013.09.003. Epub 2013 Oct 7. PMID 24144530
- [Background] Akerstedt T, Gillberg M. Subjective and objective sleepiness in the active individual. Int J Neurosci. 1990 May;52(1-2):29-37. doi: 10.3109/00207459008994241. PMID 2265922
- [Background] AMERICAN ACADEMY OF SLEEP MEDICINE 2014. International classification of sleep disorders Darien, IL: American Academy of Sleep Medicine, 3.
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] BECK, A. T., STEER, R. A. & BROWN, G.A. 1996. Manual for the Beck Depression Inventory-II. San Antonio, TX:Psychological Corporation.
- [Background] Bennett S, Alpert M, Kubulins V, Hansler RL. Use of modified spectacles and light bulbs to block blue light at night may prevent postpartum depression. Med Hypotheses. 2009 Aug;73(2):251-3. doi: 10.1016/j.mehy.2009.01.049. Epub 2009 Mar 28. PMID 19329259
- [Background] Berson DM. Phototransduction in ganglion-cell photoreceptors. Pflugers Arch. 2007 Aug;454(5):849-55. doi: 10.1007/s00424-007-0242-2. Epub 2007 Mar 10. PMID 17351786
- [Background] Brainard GC, Hanifin JP, Greeson JM, Byrne B, Glickman G, Gerner E, Rollag MD. Action spectrum for melatonin regulation in humans: evidence for a novel circadian photoreceptor. J Neurosci. 2001 Aug 15;21(16):6405-12. doi: 10.1523/JNEUROSCI.21-16-06405.2001. PMID 11487664
- [Background] Burkhart K, Phelps JR. Amber lenses to block blue light and improve sleep: a randomized trial. Chronobiol Int. 2009 Dec;26(8):1602-12. doi: 10.3109/07420520903523719. PMID 20030543
- [Background] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Dorheim SK, Bjorvatn B, Eberhard-Gran M. Insomnia and depressive symptoms in late pregnancy: a population-based study. Behav Sleep Med. 2012;10(3):152-66. doi: 10.1080/15402002.2012.660588. PMID 22742434
- [Background] Facco FL, Kramer J, Ho KH, Zee PC, Grobman WA. Sleep disturbances in pregnancy. Obstet Gynecol. 2010 Jan;115(1):77-83. doi: 10.1097/AOG.0b013e3181c4f8ec. PMID 20027038
- [Background] Gronli J, Byrkjedal IK, Bjorvatn B, Nodtvedt O, Hamre B, Pallesen S. Reading from an iPad or from a book in bed: the impact on human sleep. A randomized controlled crossover trial. Sleep Med. 2016 May;21:86-92. doi: 10.1016/j.sleep.2016.02.006. Epub 2016 Mar 2. PMID 27448477
- [Background] Hauge ER, Berle JO, Oedegaard KJ, Holsten F, Fasmer OB. Nonlinear analysis of motor activity shows differences between schizophrenia and depression: a study using Fourier analysis and sample entropy. PLoS One. 2011 Jan 28;6(1):e16291. doi: 10.1371/journal.pone.0016291. PMID 21297977
- [Background] Henriksen TE, Skrede S, Fasmer OB, Hamre B, Gronli J, Lund A. Blocking blue light during mania - markedly increased regularity of sleep and rapid improvement of symptoms: a case report. Bipolar Disord. 2014 Dec;16(8):894-8. doi: 10.1111/bdi.12265. Epub 2014 Sep 27. PMID 25264124
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Meyer TJ, Miller ML, Metzger RL, Borkovec TD. Development and validation of the Penn State Worry Questionnaire. Behav Res Ther. 1990;28(6):487-95. doi: 10.1016/0005-7967(90)90135-6. PMID 2076086
- [Background] Milton K, Bull FC, Bauman A. Reliability and validity testing of a single-item physical activity measure. Br J Sports Med. 2011 Mar;45(3):203-8. doi: 10.1136/bjsm.2009.068395. Epub 2010 May 19. PMID 20484314
- [Background] Nicassio PM, Mendlowitz DR, Fussell JJ, Petras L. The phenomenology of the pre-sleep state: the development of the pre-sleep arousal scale. Behav Res Ther. 1985;23(3):263-71. doi: 10.1016/0005-7967(85)90004-x. No abstract available. PMID 4004706
- [Background] Nodine PM, Matthews EE. Common sleep disorders: management strategies and pregnancy outcomes. J Midwifery Womens Health. 2013 Jul-Aug;58(4):368-77. doi: 10.1111/jmwh.12004. Epub 2013 Jul 15. PMID 23855316
- [Background] Pallesen S, Bjorvatn B, Nordhus IH, Sivertsen B, Hjornevik M, Morin CM. A new scale for measuring insomnia: the Bergen Insomnia Scale. Percept Mot Skills. 2008 Dec;107(3):691-706. doi: 10.2466/pms.107.3.691-706. PMID 19235401
- [Background] RØYSAMB, E., VITTERSØ, J. & TAMBS, K. 2014. The Relationship Satisfaction scale-psychometric properties. Norsk Epidemiologi, 24, 187-94.
- [Background] Sivertsen B, Omvik S, Havik OE, Pallesen S, Bjorvatn B, Nielsen GH, Straume S, Nordhus IH. A comparison of actigraphy and polysomnography in older adults treated for chronic primary insomnia. Sleep. 2006 Oct;29(10):1353-8. doi: 10.1093/sleep/29.10.1353. PMID 17068990
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Wilson DL, Barnes M, Ellett L, Permezel M, Jackson M, Crowe SF. Decreased sleep efficiency, increased wake after sleep onset and increased cortical arousals in late pregnancy. Aust N Z J Obstet Gynaecol. 2011 Feb;51(1):38-46. doi: 10.1111/j.1479-828X.2010.01252.x. Epub 2010 Dec 7. PMID 21299507
- [Derived] Liset R, Gronli J, Henriksen RE, Henriksen TEG, Nilsen RM, Pallesen S. A randomized controlled trial on the effects of blue-blocking glasses compared to partial blue-blockers on sleep outcomes in the third trimester of pregnancy. PLoS One. 2022 Jan 28;17(1):e0262799. doi: 10.1371/journal.pone.0262799. eCollection 2022. PMID 35089982
- Available data/document: Study Protocol — https://helseforskning.etikkom.no/prosjekterirek/prosjektregister/prosjekt?p_document_id=742253&p_parent_id=755398&_ikbLanguageCode=n — This is a brief description of the Project published at the web site of The Regional Ethics Committee (REC West).